CLINICAL TRIAL: NCT04320550
Title: Frequency of Functional Gastrointestinal Disorders Among School Aged Children
Brief Title: Frequency of Functional Gastrointestinal Disorders in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Ali Zohrey, Resident, Assiut University
Other Study IDs: FGIDs
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Functional Abdominal Pain Syndrome
Keywords: abdominal pain; recurrent
MeSH Terms: conditions — Abdominal Pain; Recurrence | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- abdominal pain: one group of children complaining of recurrent abdominal pain
  Interventions: Diagnostic Test: abdominal ultra sound

INTERVENTIONS:
Diagnostic Test: abdominal ultra sound — non invasive tests to exclude pathological causes
  Other Names: complete blood count; Erythrocyte sidementation rate; C reactive protein

SUMMARY:
cross sectional study to detect frequency of functional gastrointestinal disorders among schhol aged children complaining of recurrent abdominal pain

DETAILED DESCRIPTION:
school aged children from age of 5 to age of 15 who are complaining of recurrent abdominal pain will be included in the study , detailed history , examination and investigations will be done

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of recurrent abdominal pain
* the child can express and locate site of the pain

Exclusion Criteria:

* children less than 5 and adolescents more than 14
* mentally retarded children

Ages: 5 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: children with recurrent abdominal pain will be subjected to medical history , detailed examination and some investigations
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2020-12-20 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
no structural or biochemical abnormality | 1 week
  percentage of functional gastrointestinal disorders

OTHER OUTCOMES:
structural or biochemical abnormalities | 1 week
  percentage of causes of patholological recurrent abdominal pain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Reust CE, Williams A. Recurrent Abdominal Pain in Children. Am Fam Physician. 2018 Jun 15;97(12):785-793. PMID 30216016
- [Result] Chopra J, Patel N, Basude D, Gil-Zaragozano E, Paul SP. Abdominal pain-related functional gastrointestinal disorders in children. Br J Nurs. 2017 Jun 8;26(11):624-631. doi: 10.12968/bjon.2017.26.11.624. PMID 28594620